CLINICAL TRIAL: NCT01585493
Title: CHANGE.A Randomized Clinical Trial of Health Promoting Programme Versus Standard Treatment for Patients With Schizophrenia
Brief Title: CHANGE -it is About Life
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Change
Record Dates: First submitted 2012-03-27; First posted 2012-04-26 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Schizophrenia; Metabolic Syndrome
Keywords: Lifestyle; Smoking; Dietary; Exercise
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome; Smoking; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment as usual (Active Comparator): Treatment as usual
  Interventions: Other: Treatment as usual
- Care coordinator (Active Comparator)
  Interventions: Behavioral: Care coordinator
- CHANGE (Experimental)
  Interventions: Behavioral: CHANGE

INTERVENTIONS:
Other: Treatment as usual — Treatment as usual. Patients will be affiliated with local out-patient clinics in secondary mental health services and they will have access to their own general practitioner. No formalized extra effort will be made to ensure treatment of physical disorders.Patients will be affiliated with local out-patient clinics in secondary
  Arms: Treatment as usual
Behavioral: Care coordinator — Treatment as usual plus a care coordinator (with a caseload of 25 patients) who will facilitate contact to primary care in order to ensure treatment of physical health problems,
  Arms: Care coordinator
Behavioral: CHANGE — Treatment as usual plus affiliation to a staffmember (caseload 10) from a CHANGE team who will provide individualized, adjusted implementation of widely recognized interventions, such as smoking cessation programmes, motivational interviewing, psychoeducation plus patient involvement in monitoring health statusA multidisciplinary CHANGE team will be established. Team members will be health professionals with experience in smoking cessation programmes or exercise programmes for mentally ill, and experts with competence in dietary issues.
  CHANGE treatment involve lifestyle coaching, education about diet and physical activity,16 networking and smoking cessation programs. The team members will act as lifestyle coaches for ten patients at a time, map lifestyle and explore and elicit patients' motivation for change.
  Arms: CHANGE

SUMMARY:
Schizophrenia is a life shortening disease, not only because of suicide but also because of increased mortality from natural causes. Recently, a large register-based study, involving complete national data from Denmark, Sweden and Finland, showed that life expectancy for schizophrenia is 20 years shorter for men and 15 years shorter for women, compared to the general population, and that mortality from medical conditions and diseases are responsible for a large proportion of the reduced life expectancy. Patients with schizophrenia had a twofold to fivefold increased risk of death by coronary heart disease, respiratory diseases, lung cancer and metabolic conditions. Unhealthy life style and undetected and untreated physical disorders play an important role in this excess mortality.Results from the Danish National Indicator Project for Schizophrenia showed that a much higher proportion of patients with schizophrenia compared to the general population have measures of waist circumference, body mass index, blood pressure, blood lipids and blood glucoses above the recommended upper values.

In the randomized clinical trial CHANGE, the investigators will evaluate the effect of two different interventions both aiming to reduce risk for death from medical diseases. We will compare 1) treatment as usual with 2) affiliation to a care coordinator who has the duty to connect the patient to general practice and primary care and 3) affiliation to a staff member from the CHANGE team who should facilitate life style changes and contact with general practice. The objective is to identify interventions that can reduce the risk of early death in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to outpatients services at Mental Health Centre, Copenhagen or Århus University Hospital
* Diagnose ICD-10:F2 spectrum
* Waist circumference > 88 cm for women or >102 cm for men

Exclusion Criteria:

* Not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2012-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Copenhagen Risk Score | 12 months
  The primary outcome is change in 10 years risk of cardiovascular disease from baseline at 12 months.

SECONDARY OUTCOMES:
Smoking | 12 months
  Number of daily smokers in each group at 12 months
Sedentary lifestyle | 12
  Self reported hours of sedentary behavior
Body mass index | 12 months
  Change in body mass index at 12 months
Blood pressure | 12 months
  Change in systolic and diastolic blood pressure at 12 months
Cholesterol | 12 months
  Change in total Cholesterol, LDL, HDL, and triglycerides and 12 months
Aerobic fitness | 12 months
  Indirectly estimated maximal oxygen uptake
Waist circumference | 12 months
  Measured between crista iliaca and the lowest rib
Forced expiratory volume | 12 months
Resting heart rate | 12 months
HbA1c | 12 months
Physical activity | 12 months
  Change in minutes of MVPA a week

OTHER OUTCOMES:
Positive and negative symptoms | 12 months
Cognition | 12 months
Quality of life | 12 months
Dietary pattern | 12 months
Self rated health | 12 months
High sensitive CRP | 12 months
Triglycerides | 12 months
Global assessment functioning (GAF) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Merete Nordentoft, Professor, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (1):
- Mental Health Services in the Capital Region, Denmark, Copenhagen, Denmark

REFERENCES:
- [Derived] Speyer H, Norgaard HC, Hjorthoj C, Madsen TA, Drivsholm S, Pisinger C, Gluud C, Mors O, Krogh J, Nordentoft M. Protocol for CHANGE: a randomized clinical trial assessing lifestyle coaching plus care coordination versus care coordination alone versus treatment as usual to reduce risks of cardiovascular disease in adults with schizophrenia and abdominal obesity. BMC Psychiatry. 2015 May 23;15:119. doi: 10.1186/s12888-015-0465-2. PMID 26001844